CLINICAL TRIAL: NCT06843915
Title: Aerobic Exercise as a Therapeutic Approach for Urinary Incon-tinence in Multiple Sclerosis: Insights From a Pilot Randomized Controlled Trial
Brief Title: Aerobic Exercise for Urinary Incontinence in Multiple Sclerosis
Acronym: UI-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Alham Al-Sharman, Associate prof, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUST-AA-2015-182
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis; Urinary Incontinence
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Aerobic Exercise group (MIAE) (Experimental): Participants in the moderate-intensity aerobic exercise (MIAE) group engaged in a 40-minute supervised session using the StepOne-SCIFIT recumbent stepper machine. The session included a 5-minute warm-up at 25 watts, followed by 30 minutes of moderate-intensity exercise, main-taining a stepping rate of 90-100 steps per minute. The workload was adjusted to keep the participant's heart rate within the target heart rate range (THRR), calculated using the Karvonen formula. During the first three weeks, the exercise intensity was set at 50-59% of heart rate reserve (HRR), and for the remaining three weeks, it was increased to 60-69% of HRR. Polar heart rate monitors were used to assess heart rate before and after each session. Participants kept weekly exercise logs to monitor compliance.
  Interventions: Other: Moderate intensity aerobic exercise
- Home Exercise Program group (HEP) (Active Comparator): Participants in the home exercise program (HEP) group received a Digital video disc (DVD) exercise and a printed manual covering low-intensity, non-aerobic exercises to control for general activity levels. The DVD, developed for individuals with movement disorders, was in Arabic and included warm-up and cool-down activities, flexibility, strength, balance, endurance exercises, and relaxation techniques. The examiner reviewed the DVD and precautions with each participant to ensure correct execution. Participants were also monitored for adherence through weekly exercise logs.
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Other: Moderate intensity aerobic exercise — Participants in the MIAE group engaged in a 40-minute supervised session using the StepOne-SCIFIT recumbent stepper machine. The session included a 5-minute warm-up at 25 watts, followed by 30 minutes of moderate-intensity exercise, main-taining a stepping rate of 90-100 steps per minute. The workload was adjusted to keep the participant's heart rate within the target heart rate range (THRR), calculated using the Karvonen formula. During the first three weeks, the exercise intensity was set at 50-59% of heart rate reserve (HRR), and for the remaining three weeks, it was increased to 60-69% of HRR. Polar heart rate monitors were used to assess heart rate before and after each session. Participants kept weekly exercise logs to monitor compliance.
  Arms: Moderate-Intensity Aerobic Exercise group (MIAE)
Other: Home Exercise Program — Home Exercise Program
  Arms: Home Exercise Program group (HEP)

SUMMARY:
Limited studies has investigated the effect of aerobic exercise program on urinary inconitenance in people with multiple sclerosis. This study aims to explore the effects of a six weeks moderate-intensity aerobic exercise intervention on UI and UI related bi-omarkers specifically cortisol using. Urinary incontinence and blood samples were assessed after 6-week intervention of aerobic exercise.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a prevalent and debilitating issue in people with Multiple Sclerosis (PwMS). This condition reduces the quality of life for those affected by MS, imposing substantial physical, emotional, and social burdens. Certainly, emphasizing the necessity for effective UI management strategies in the context of MS. Physical activity was associated with a significant reduction in urinary incontinence. Aerobic exercise, commonly referred to as "cardio," improves the heart's efficiency in pumping oxygenated blood, thus supplying essential oxygen to active muscles.

During aerobic exercise, stabilizing muscles such as the abdominals and adductors are significantly engaged. Given that Pelvic floor muscles (PFMs) are critical for the voluntary urinary continence mechanism, they also serve as stabilizers and postural muscles, capable of reflexive activation during physical activity. Therefore, PFMs are essential for maintaining continence and providing effective pelvic stabilization. Recent systematic review has found that there is moderate evidence that the aerobic and/or resistance exercise program associated with PFM training compared to usual care can reduce UI in pregnant women.

This pilot study utilized a single-blinded, randomized controlled design to estab-lish the groundwork for calculating effect sizes for future Phase II randomized con-trolled trials (RCTs), following Hertzog's (2008) guidelines. The study compared two groups: an intervention group participating in a six-week moderate-intensity aerobic exercise program, and a control group engaged in non-aerobic exercises at home.

Participants were recruited from patients with MS attending routine neurology appointments at King Abdullah University Hospital (KAUH-Irbid, Jordan) between November 2018 and May 2020. Initial eligibility screening was conducted, and eligible patients were invited to participate. Patients who had previously consented to be contacted for future research or had participated in other studies were also approached. Information about the study was shared via the Jordanian Multiple Sclerosis Society, and interested patients underwent further eligibility screening.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis by a neurologist based on the revised McDonald criteria.
* Expanded Disability Status Scale (EDSS) score between 3 and 5.5
* No symptom exacerbation in the 30 days before testing
* Aged 18 years or older
* Ability to provide informed consent
* Absence of urinary incontinence (UI) before MS onset
* no history of pelvic surgery, radiotherapy, or bladder stones.

Exclusion Criteria:

* Inability to perform the exercise test on a recumbent stepper
* Recent acute ischemic cardiovascular event or coronary artery bypass surgery within the past three months
* severe uncorrected visual impairments
* Uncontrolled hy-pertension (blood pressure > 190/110 mmHg) despite medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Incontinence Questionnaire short-form ques-tionnaire (ICIQ-UI SF) | 6 Weeks
  The International Consultation on Incontinence Questionnaire short-form ques-tionnaire (ICIQ-UI SF) was used to assess the presence and frequency of UI in our pa-tient cohort. The questionnaire has been validated and widely used in clinical and re-search settings to evaluate urinary symptoms and quality of life. It serves as a valuable tool for healthcare providers and researchers in evaluating the prevalence, frequency, severity, and the impact of UI on the quality of life (QoL) of individuals affected by this neurological condition as per MS. The Arabic version of the ICIQ_UI_SF was used in this study. The total ICIQ-UI SF score ranges from 0 to 21 points, with the severity being classified according to the total score: 0-7 points for mild UI, 8-12 points for moderate UI, and 13-21 points for severe UI.

SECONDARY OUTCOMES:
Plasma Cortisol level | 6 Weeks
  Blood samples were collected for measurement of cortisol from MS participants in both groups at 8:00 am ±1 hour to standardize for daily physiological variations in cor-tisol. Cortisol determinations was examined using competitive enzyme-linked im-mune-sorbent assay technology while Serum/plasma serotonin level was examined using Sandwich enzyme-sorbent assay technology. After blood collection, all blood samples were centrifuged at 1500 x g for 15 minutes in order to collect serum. Following to this, serums were stored at -80°C until used. A competitive ELISA kits for quantita-tive analysis of total serum cortisol was used. All assays were performed according to the instructions provided by the manufacturer.

CONTACTS AND LOCATIONS:
Locations (1):
- Naseem Oudah, Irbid, Jordan